CLINICAL TRIAL: NCT03486418
Title: Development of an Endoscopic Classification Score System for Serrated Adenomas in the Colorectum
Brief Title: European Serrated Adenoma Classification Score
Acronym: ESCO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: ESCO
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Colorectal polyps
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to develop a score system in order to differentiate adenomatous polyps, hyperplastic polyps and serrated adenomas on the basis of optical features. Endoscopic images of colorectal polyps will be collected from a prospectively managed database. Histopathological diagnoses are available for all polyps. Histopathological diagnoses serve as gold standard in this study.

In the first phase of the study optical features of serrated adenomas are extracted from the database. Discriminators are then defined on the basis of the extracted features. In the second phase a test set of high quality pictures are provided to both novices and experts of colorectal endoscopy. Participants are asked to use the above named discriminators in order to rate pictures and to classify polyps into three classes (adenomatous polyps, hyperplastic polyps and serrated adenomas). In the third phase of the study accuracy of optical bases diagnoses is calculated by comparing optically derived diagnoses with histopathological diagnoses (gold standard).

ELIGIBILITY:
Inclusion Criteria:

* indication for colonoscopy
* patients >= 18 years

Exclusion Criteria:

* pregnant women
* indication for colonoscopy: inflammatory bowel disease
* indication for colonoscopy: polyposis syndrome
* indication for colonoscopy: emergency colonoscopy e.g. acute bleeding
* contraindication for polyp resection e.g. patients on warfarin

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Optical diagnosis of each colorectal polyp | Participants will be followed for the duration of the study an expected average of 6 month
  The predicted polyp histology (determined according to optical polyp features) will be assessed; the predicted diagnosis will be compared with the histopathological diagnosis (gold standard) after;

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum rechts der Isar der TU München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No